CLINICAL TRIAL: NCT06424717
Title: A Single Arm, Open-label, Multicenter, Phase 2 Study to Evaluate the Efficacy, Safety, and Tolerability of Avelumab in Combination With the ATR Inhibitor Tuvusertib in Participants With Advanced Urothelial Carcinoma That Has Progressed on Prior Anti-PD-(L)1 Therapy (JAVELIN DDRiver Bladder)
Brief Title: Study of Avelumab and Tuvusertib in Participants With Advanced Urothelial Cancer That Has Progressed on Prior Anti-PD-(L)1 Therapy (JAVELIN DDRiver Bladder)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial withdrawn based on re-prioritization of the clinical development path for tuvusertib. No subjects were enrolled.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS202611_0001; 2024-511203-42-00 (Other: EU CT Number)
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Urothelial Carcinoma
Keywords: M1774; locally advanced and unresectable or metastatic urothelial carcinoma; bladder cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab with tuvusertib (Experimental)
  Interventions: Drug: Avelumab; Drug: Tuvusertib

INTERVENTIONS:
Drug: Avelumab — Participants will be administered Avelumab intravenously (IV).
  Other Names: MSB0010718C
Drug: Tuvusertib — Participants will be administered Tuvusertib orally.
  Other Names: M1774

SUMMARY:
The purpose of this study is to assess the antitumor activity of avelumab in combination with tuvusertib in terms of objective response in participants with advanced urothelial carcinoma. Study details include:

Condition/Disease: Participants with urothelial carcinoma (locally advanced and unresectable, or metastatic) that has progressed on prior anti-PD-(L)1 therapy Treatment Duration: Participants will be treated until progressive disease, death, or discontinuation due to e.g. withdrawal of consent or lost to follow-up Visit Frequency: While receiving study intervention, participants will visit the site twice per every 21-day study intervention period. 1 week after end of study intervention, participants will visit the site for an End of Study Intervention Visit, followed by 2 Safety Follow-Up visits at 1 and 3 months after last dose, and thereafter have remote Long-Term Follow-up every 3 months.

Study Duration: The overall study is planned to close after the last participant has been followed up for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally advanced, and unresectable or metastatic urothelial carcinoma.
* No more than 2 lines of therapy for advanced disease. Chemotherapy followed by avelumab (switch maintenance) counts as 1 line of therapy. Additionally, (neo)-adjuvant chemotherapy for Muscle invasive bladder cancer with recurrence or progression within 12 months of last dose, counts as a line of therapy.
* Measurable disease by RECIST 1.1, as assessed by the Investigator.
* Eastern Cooperative Oncology Group Performance status 0 to 1.
* Adequate hematologic function as indicated by:
* Platelet count more than or equal to 100,000 per microliter
* Absolute neutrophil count more than or equal to 1,500 per microliter with no growth factor treatment within the last 14 days
* Hemoglobin more than or equal to 9.0 gram/deciliter with no erythropoietin or red blood cell transfusion within the last 14 days
* Only one line of an antibody-drug conjugate (ADC) is allowed.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Any condition, including any uncontrolled disease state other than aUC, that in the Investigator's opinion constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation.
* Any known additional malignancy that is progressing and/or requires active treatment including adjuvant hormonal therapy.
* Presence of brain metastases unless clinically stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of study intervention and any neurologic symptoms have returned to baseline and sequelae that are a consequence of the treatment of the brain metastases are acceptable), no evidence of new brain metastases, and on a stable or decreasing dose or without steroids for at least 14 days prior to first dose of study intervention. Participants with carcinomatous meningitis are excluded regardless of clinical stability.
* Serious gastrointestinal bleeding within 3 months, refractory nausea and vomiting, uncontrolled diarrhea, known malabsorption, significant small bowel resection or gastric bypass surgery, use of feeding tubes, other chronic gastrointestinal disease (including exocrine pancreatic insufficiency requiring pancreatic enzyme replacement therapy), and/or other situations that may preclude adequate absorption of oral medications.
* Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-16 (Estimated); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
Confirmed Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors(RECIST) v1.1 as Assessed by Investigator in Participants with Selected Tumor Chromatin Modifier Mutations | Up to 18 months

SECONDARY OUTCOMES:
Confirmed Objective Response (OR) According to RECIST v1.1 as Assessed by Investigator | Up to 18 months
Duration of Response (DoR) According to RECIST 1.1 as Assessed by the Investigator | Up to 18 months
Progression Free Survival (PFS) According to RECIST 1.1 as Assessed by the Investigator | Up to 18 months
Overall Survival (OS) | From the date of randomization until death, assessed up to 1.5 years
Number of Participants With Treatment-Emergent Adverse Events (TEAE), Serious TEAEs and Related TEAEs | Up to 18 months
Confirmed Objective Response (OR) According to RECIST v1.1 as Assessed by Investigator in Subpopulations as Defined by Selected Tumor Biomarkers | Up to 18 months
Duration of Response (DoR) According to RECIST 1.1 as Assessed by the Investigator in Subpopulations as Defined by Selected Tumor Biomarkers | Up to 18 months
Progression Free Survival (PFS) According to RECIST 1.1 as Assessed by the Investigator in Subpopulations as Defined by Selected Tumor Biomarkers | Up to 18 months
Overall Survival (OS) in Subpopulations as Defined by Selected Tumor Biomarkers | From the date of randomization until death, assessed up to 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html